CLINICAL TRIAL: NCT06223100
Title: An Observational Study on the Efficacy and Safety of the Combination Regimen Based on Eravacycline in the Treatment of Multidrug-resistant Bacterial Infections in Immunocompromised Host Populations.
Brief Title: Efficacy and Safety of the Combination Therapy Based on Eravacycline in Immunocompromised Hosts With MDROS Infection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lingai Pan, Associate Clinical Professor, Sichuan Provincial People's Hospital
Other Study IDs: LPan20230578
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Immune Dysregulation Disorder
MeSH Terms: interventions — eravacycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Abdominal drainage fluid samples, blood samples, respiratory tract samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Eravacycline — There is no other intervention.
  Other Names: XERAVA

SUMMARY:
The goal of this observational study is to explore the treatment mode and clinical outcome of patients with immunocompromised who received the combined regimen of eraracycline in the treatment of multidrug-resistant bacterial infections, to evaluate the efficacy and safety of the combined regimen of eravacycline in the treatment of multidrug-resistant bacterial infections in immunocompromised host populations, and to provide data reference for the treatment of immunocompromised populations.

DETAILED DESCRIPTION:
The goal of this observational study is to explore the treatment mode and clinical outcome of patients with immunocompromised who received the combined regimen of eraracycline in the treatment of multidrug-resistant bacterial infections, to evaluate the efficacy and safety of the combined regimen of eravacycline in the treatment of multidrug-resistant bacterial infections in immunocompromised host populations, and to provide data reference for the treatment of immunocompromised populations. The main questions it aims to answer are:

* The 30-day all-cause mortality of multi-drug resistant bacterial infections in immunocompromised host populations treated with the combined regimen of eravacycline ;
* Evaluate the clinical cure rate and symptom improvement rate of eravacycline treatment.

According to the clinical practice (symptoms, signs, imaging, culture and drug sensitivity, etc.), the doctor determines the combined regimen of eravacycline, and the combined drugs are used routinely according to their instructions or clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old.
* Voluntary to participate in this study and signed informed consent. If the subject is unable to read and / or sign the informed consent due to incapacity or other reasons, the guardian of the subject is required to act as the agent of the informed process and sign the informed consent.
* In a state of low immune function:
* In this study, if the patient meets any of the following criteria, the patient 's immune function is considered to be low : 1 patients who have previously received solid organ transplantation ( liver, kidney, lung, heart ) ; 2 hematological malignancies ( leukemia, lymphoma ) ; 3 Patients received long-term immunosuppressive therapy, or used steroids that reached immunosuppressive doses within 21 months before screening ( ≥ 10 mg prednisone or > 15 mg / kg / d hydrocortisone or d > 3 mg / kg / d methylprednisolone, continuous d > 5 days ) [ 4,13 ]. 4 Severe infections occurred recently, leading to extremely low immune function.
* Infections caused by known or highly suspected multidrug-resistant pathogens (MDR), or gram-negative bacteria that are sensitive to eravacycline in adult patients with limited treatment options. The high-risk factors and standards of MDR met the definition of " Chinese expert consensus on prevention and control of nosocomial infection of multidrug-resistant bacteria "; multidrug-resistant bacteria (MDR) refer to bacteria that are resistant to three or more types of commonly used antibiotics that are usually sensitive. Multidrug resistance also includes pan-drug resistance (XDR) and pan-drug resistance (PDR).
* Patients treated with elastin ≥ 3 days.

Exclusion Criteria:

* Urinary tract infection.
* Clear culture results showed that microbial pathogens were not sensitive to test drugs (such as Pseudomonas aeruginosa, etc.).
* Patients whose expected survival time cannot exceed the study period.
* The researchers believe that there is any medical history, current condition, treatment, abnormal laboratory examination or other conditions that may affect the test results, interrupt the test process (or the subject cannot complete all the operations and visits required by the test) or accept the test drugs that will increase the risk of the subject. Patients with end-stage diseases have immediate life-threatening disease evidence.
* Patients with a history of allergic reactions to tetracyclines or any adjuvant contained in the study drug formula.
* Vulnerable groups other than critically ill patients, including people with mental illness, cognitive impairment, pregnant women, etc.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with low immune function are at high risk of multidrug-resistant bacterial infections, especially those who need long-term immunosuppressive therapy, such as patients with hematological malignancies, solid organ transplant recipients, etc.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause mortality | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  Evaluate the 30-day all-cause mortality of multi-drug resistant bacterial infections in immunocompromised host populations treated with the combined regimen of eravacycline.
Clinical cure rate | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  Evaluate the clinical cure rate of eravacycline treatment.
Symptom improvement rate | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  Evaluate the symptom improvement rate of eravacycline treatment.

SECONDARY OUTCOMES:
Safety and tolerance of eravacycline | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  Safety evaluation was mainly based on the incidence of adverse events / adverse reactions in the two groups of patients.
Microbial clearance rate | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  In patients who met all clinical evaluation criteria and had positive bacterial culture before treatment, the microbiological efficacy was evaluated at the end of treatment and after treatment (discharge). The results of follow-up (discharge) after treatment were the main evaluation endpoints, and the bacterial clearance rate was calculated. The microbiological efficacy was determined according to the following criteria: clearance, assumed clearance, non-clearance, assumed non-clearance, partial clearance, and others.
Impact of different treatment timing on eravacycline outcomes as assessed by 30-day all-cause mortality. | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  The timing of treatment refers to the time when the patients with positive previous culture results start the treatment with eravacycline, one of which assessed the 30-day all-cause mortality of multi-drug resistant bacterial infections in immunocompromised host populations treated with the combined regimen of eravacycline.
Impact of different treatment timing on eravacycline outcomes as assessed by clinical cure rates. | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  The timing of treatment refers to the time when the patients with positive previous culture results start the treatment with eravacycline, one of which assessed the clinical cure rate of eravacycline treatment.
Impact of different treatment timing on eravacycline outcomes as assessed by clinical improvement rates. | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  The timing of treatment refers to the time when the patients with positive previous culture results start the treatment with eravacycline, one of which assessed the symptom improvement rate of eravacycline treatment.
The 30-day infection recurrence rate | during the treatment (1-14 days); the end of treatment（Day 14）; 28-35 days after first dose
  The 30-day infection recurrence rate